CLINICAL TRIAL: NCT02574052
Title: Medical College Students' Responds to Menu Labeling With or Without Nutrition
Brief Title: Medical College Students' Responds to Menu Labeling
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Kaimeng Kong, Department of Clinical Nutrition, Xinhua Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, China, Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XHEC-C-2014-094
Record Dates: First submitted 2015-10-07; First posted 2015-10-12 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-10

CONDITIONS: Dietary Modification
Keywords: Menu Labelling;; Nutrition Education;; dietary assessment tools;
MeSH Terms: interventions — Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Behavioral (Other): The whole experiment was divided into three phases with each phase lasting two weeks.
  First Stage-Behavioral: just record participants' food choices Second Stage-Behavioral: menu labelling without nutrition education Third Stage- Behavioral; menu labelling with nutrition education
  Interventions: Behavioral: participants' food choices; Behavioral: menu labelling without nutrition education; Behavioral: menu labelling with nutrition education

INTERVENTIONS:
Behavioral: participants' food choices — just recorded the participants' food choices in the school cafeteria
Behavioral: menu labelling without nutrition education — The investigators provided every participant with a menu labeling without any interpretation and recorded their dietary selections
Behavioral: menu labelling with nutrition education — The investigators not only sent a menu labeling to every participant, but also delivered nutrition education to participants by providing them with nutrition and health knowledge through WeChat daily.

SUMMARY:
The purpose of this study is to evaluate whether exposure to nutrition information with or without nutrition education would influence college students' dietary choices and improved the previous photographs-based dietary assessment tools.

DETAILED DESCRIPTION:
1. The investigators improved the previous photographs-based dietary assessment tools and utilized the improved approach to evaluate participants' calorie and nutrients intake.
2. A pre-post non-controlled study design was implemented in the medical college and was divided into three stages: just recording the dietary selection in the three meals daily, recording the dietary selection with the provision of menu labeling accompanying with or without nutrition education. The investigators adopted photographs-based dietary assessment tools and a mobile phone application 'WeChat' was utilized as the photographs and nutrition knowledge transfer platform. Two professional researchers respectively read the received photographs and calculated participants' calorie and nutrients intake.

ELIGIBILITY:
Inclusion Criteria:

* Grade 2012, 2013 undergraduate students and Grade 2013 graduate students

Exclusion Criteria:

* Participants who sent the photographs less than six times in any one of the three meals at any stage

  * Participants who did not complete their questionnaires

    * Participants who withdrew from the experiment at any stage

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2014-10; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Descriptive Name of Scale: Composite outcome measure of calorie (kcal/day), protein(g/day), fat intake (g/day) and carbohydrate intake (g/day) of participants | up to six weeks
  Through the receiving photographs the participants took about their three meals, the investigators estimated the calorie content (kcal/day), protein content (g/day), fat content (g/day), carbohydrate content (g/day) participants ate.

CONTACTS AND LOCATIONS:
Overall Officials: Yexuan Tao, PH.D, M.D, Principal Investigator — Xinhua Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, China

REFERENCES:
- [Background] Chu YH, Frongillo EA, Jones SJ, Kaye GL. Improving patrons' meal selections through the use of point-of-selection nutrition labels. Am J Public Health. 2009 Nov;99(11):2001-5. doi: 10.2105/AJPH.2008.153205. Epub 2009 Sep 17. PMID 19762664
- [Background] Harnack LJ, French SA, Oakes JM, Story MT, Jeffery RW, Rydell SA. Effects of calorie labeling and value size pricing on fast food meal choices: results from an experimental trial. Int J Behav Nutr Phys Act. 2008 Dec 5;5:63. doi: 10.1186/1479-5868-5-63. PMID 19061510
- [Background] Elbel B, Gyamfi J, Kersh R. Child and adolescent fast-food choice and the influence of calorie labeling: a natural experiment. Int J Obes (Lond). 2011 Apr;35(4):493-500. doi: 10.1038/ijo.2011.4. Epub 2011 Feb 15. PMID 21326209
- [Background] Finkelstein EA, Strombotne KL, Chan NL, Krieger J. Mandatory menu labeling in one fast-food chain in King County, Washington. Am J Prev Med. 2011 Feb;40(2):122-7. doi: 10.1016/j.amepre.2010.10.019. PMID 21238859
- [Background] Sinclair SE, Cooper M, Mansfield ED. The influence of menu labeling on calories selected or consumed: a systematic review and meta-analysis. J Acad Nutr Diet. 2014 Sep;114(9):1375-1388.e15. doi: 10.1016/j.jand.2014.05.014. Epub 2014 Jul 16. PMID 25037558
- [Background] Conklin MT, Cranage DA, Lambert CU. College students' use of point of selection nutrition information. Top Clin Nutr 2005;20:97-108.
- [Background] Huybregts L, Roberfroid D, Lachat C, Van Camp J, Kolsteren P. Validity of photographs for food portion estimation in a rural West African setting. Public Health Nutr. 2008 Jun;11(6):581-7. doi: 10.1017/S1368980007000870. Epub 2007 Aug 9. PMID 17686204
- [Background] Lazarte CE, Encinas ME, Alegre C, Granfeldt Y. Validation of digital photographs, as a tool in 24-h recall, for the improvement of dietary assessment among rural populations in developing countries. Nutr J. 2012 Aug 29;11:61. doi: 10.1186/1475-2891-11-61. PMID 22931128
- [Background] Martin CK, Correa JB, Han H, Allen HR, Rood JC, Champagne CM, Gunturk BK, Bray GA. Validity of the Remote Food Photography Method (RFPM) for estimating energy and nutrient intake in near real-time. Obesity (Silver Spring). 2012 Apr;20(4):891-9. doi: 10.1038/oby.2011.344. Epub 2011 Dec 1. PMID 22134199
- [Result] Farley TA, Caffarelli A, Bassett MT, Silver L, Frieden TR. New York City's fight over calorie labeling. Health Aff (Millwood). 2009 Nov-Dec;28(6):w1098-109. doi: 10.1377/hlthaff.28.6.w1098. Epub 2009 Oct 6. PMID 19808704
- [Result] Roberto CA, Larsen PD, Agnew H, Baik J, Brownell KD. Evaluating the impact of menu labeling on food choices and intake. Am J Public Health. 2010 Feb;100(2):312-8. doi: 10.2105/AJPH.2009.160226. Epub 2009 Dec 17. PMID 20019307